CLINICAL TRIAL: NCT03910582
Title: A Randomized Clinical Trial of Endometrial Histological Dating for Personalized Frozen-thawed Embryo Transfer (pFET) in Patients With Repeated Implantation Failure (RIF) in Natural Cycle
Brief Title: Personalized FET in RIF Patients With Displaced Dating
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2019003
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subjects in this group will be treated with personalized frozen-thawed embryo transfer. The blastocysts were delayed or advanced transferred after ovulation depending on the endometrium dating in RIF group
  Interventions: Procedure: personalized frozen-thawed embryo transfer
- Control group (Active Comparator): Subjects in this group will be treated with routine frozen-thawed embryo transfer.The blastocysts were transferred 5 days after ovulation regardless of endometrium dating in control group.
  Interventions: Procedure: routine frozen-thawed embryo transfer

INTERVENTIONS:
Procedure: personalized frozen-thawed embryo transfer — The blastocysts were delayed or advanced transferred after ovulation depending on the endometrium dating in RIF group
  Arms: Experimental group
Procedure: routine frozen-thawed embryo transfer — The blastocysts were transferred 5 days after ovulation regardless of endometrium dating in control group.
  Arms: Control group

SUMMARY:
The endometrium becomes receptive as a result of a series of timed hormonal events during the menstrual cycle. The exposure of the endometrium to progesterone after ovulation initiates morphological and functional alterations that result in the change from a pre-receptive to a receptive endometrium. The morphological changes observed on histology for each specific day after ovulation were described by Noyes and his colleagues in 1950. An endometrial biopsy that shows a difference of more than 2 days between the histologic dating and actual day after ovulation is considered to be "out of phase" However, the clinical application of the Noyes criterion is relatively limited. We have verified the Noyes criterion in natural cycle in previous study which conducting endometrial biopsies respectively on day 3, 5, 7, 9 and 11 of post-ovulation (PO+3/5/7/9/11)(unpublished data).

The clinical value of the endometrial histological dating in RIF patients in natural cycle is still to be answered. In this study, we tried to investigate the clinical effects of pFET in unexplained RIF patients according to the use of classic histologic endometrial dating to estimate the timing of the window of implantation and to adjust embryo transfer time in natural cycle.

ELIGIBILITY:
Inclusion Criteria:

1. RIF patients (RIF is defined as the absence of a gestational sac on ultrasound at 5 or more weeks after 3 embryo transfers with high quality embryos or after the transfer of ≥10 embryos in multiple transfers);
2. Out of phase dating patients;
3. FET in natural cycle;
4. Single blastocysts embryo transfer;

Exclusion Criteria:

1. uterine abnormalities (double uterus, bicornuate uterus, unicornuate uterus and uterine mediastinum), intrauterine adhesions, endometriosis,adenomyosis, hydrosalpinx, and uterine fibroids (submucosal fibroids, non-mucosal fibroids> 4 cm and/or endometrial pressure);

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-04-10 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
ongoing clinical rate | 6 weeks
  Ongoing pregnancy was defined as at least one intrauterine gestational sac with cardiac action by ultrasound performed 6 weeks after ET.

SECONDARY OUTCOMES:
implantation rate | 2 weeks
clinical pregnancy rate | 4 weeks
early abortion rate | 6 weeks